CLINICAL TRIAL: NCT04413240
Title: Clinical Efficacy and Cost-effectiveness of Telerehabilitation for Post-stroke Patients
Brief Title: Telerehabilitation for Post-stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: IRCCS San Camillo, Venezia, Italy (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Chief of the Neurorehabilitation Unit. Full Professor., Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Finalizzata RF-2016-02363044
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Stroke Sequelae
Keywords: Healthcare organizations; Integrated care delivery systems; Cost-benefit analysis; Stroke; Pharmacoeconomics; Rehabilitation; Telerehabilitation; Healthcare organizations, programs, and delivery of services; Disease management and modeling
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: A clinical study with medical device, multicenter, single-blind, randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Patients in this group will undergo 20 sessions (1 hour a day, 5 days a week for 4 consecutive weeks) of "multidomain" telerehabilitation (motor, speech and/or cognitive) with VRRS, K-Wand and Khymu connected to a workstation (Telecockpit).
  Interventions: Device: Telerehabilitation
- Conventional rehabilitation group (Active Comparator): The patients assigned to this group will undergo 20 sessions (1 hour a day, 5 days a week for 4 consecutive weeks) of "multidomain" rehabilitation (motor, speech and/or cognitive). It is not possible a priori to precisely define the instruments that will be used during rehabilitation management. The telerehabilitation or conventional treatment methods (type of therapeutic exercise, modality of cognitive stimulation and/or taking care of speech therapy) will be determined for each patient on the basis of the needs emerging from the physiatric examination performed at T0, defined according to the Individual Rehabilitation Project and applied according to each Rehabilitation Program (motor, cognitive and/or speech therapy) periodically updated.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Telerehabilitation — * VRRS is a medical device to perform cognitive telerehabilitation and home speech therapy in online or offline mode.
  * K-Wand is an additional device to VRRS for motor telerehabilitation of the upper limb and trunk. It works with a set of motion sensors through light recognition technology.
  * Khymu is a set of sensors added to the VRRS used to carry out motor telerehabilitation activities of the lower limb. The use in combination with the K-Wand is able to allow "full-body" motor telerehabilitation.
  Patients will have at their home a special workstation connected to the internet. The same equipment will also be present in the reference structure. Only the online telerehabilitation mode will be used, including an audio and video teleconference. The rehabilitator will be able to remotely control the patient's system. The patient, will see on his screen the exercises to be performed, their realization and the results achieved.
  Arms: Telerehabilitation group
Other: Conventional rehabilitation — It is not possible a priori to precisely define the instruments that will be used during rehabilitation management. The telerehabilitation or conventional treatment methods (type of therapeutic exercise, modality of cognitive stimulation and/or taking care of speech therapy) will be determined for each patient on the basis of the needs emerging from the physiatric examination performed at T0, defined according to the Individual Rehabilitation Project and applied according to each Rehabilitation Program (motor, cognitive and/or speech therapy) periodically updated.
  Arms: Conventional rehabilitation group

SUMMARY:
In the last few years, there has been an increasing shift towards outpatients setting in the care of patients with stroke. Unfortunately, this led to a high percentage of discharged patients who did not receive an adequate amount of rehabilitation, because of some non-clinical factors, such as resource availability, geographical location, age, and personal wealth. To date, there is growing evidence about the role of telerehabilitation as an effective method to deliver rehabilitative treatments to homebound subjects with no moving of therapists or patients. However, the most appropriate organizational models regarding Health Technology Assessment in telerehabilitation procedures still object of debate. On these bases, the aim of this project is to investigate the feasibility and effectiveness of multi-domains telerehabilitation procedures in stroke patients in order to supply the National Health Service with some useful information about the use of telerehabilitation in clinical practice of stroke rehabilitation.

DETAILED DESCRIPTION:
In the last few years, due to limited resources, stroke patients hospitalization has been progressively shortened with the increasing shift of some rehabilitation procedures towards outpatient settings. This led to a high percentage of discharged patients who doesn't receive an adequate amount of rehabilitation. This was because of some non-clinical factors, such as resources availability, geographical location, age and personal wealth. Unfortunately, the benefits gained during inpatient rehabilitation are often not sustained in the long term. Thus stroke patients progressively decrease their activity level leading to functional deterioration. To face these difficulties, telerehabilitation may be useful to deliver rehabilitative treatments to homebound subjects with no moving of therapists or patients. To date some studies highlighted that rehabilitation delivered from-distance has similar results of face-to-face one, confirming that telerehabilitation may be effectively used to address the growing call for improving home care. Despite these observations, telerehabilitation is still few integrated into outpatients territorial rehabilitative practice. Furthermore, the current literature about telerehabilitation is mainly focused on a single domain of intervention (i.e. motor, cognitive, speech), with scant data about the impact of telerehabilitation on global disability. Finally, the cost-benefit ratio of telerehabilitation, compared to usual territorial rehabilitation or prolonged hospitalization, still objects of debate.

Preliminary Data:

Previous literature about telerehabilitation evidenced an improved upper limb motor function with positive interaction stroke patient-therapist. A previous RCT evidenced similar recovery of motor performances in stroke patients who received telerehabilitation compared to "face to face" treatment. Moreover, was highlighted that patients treated with telerehabilitation were able to have good management of the system and a good relationship with therapists. Recently was showed feasibility and effectiveness of speech telerehabilitation, applied to lexical deficits in chronic stroke patients as well as of cognitive telerehabilitation in people with mild cognitive impairment, with results similar to "face-to-face" treatment.

In a systematic review on motor telerehabilitation, was supported the equivalence of "face to face" and "from a distance" delivery of neuromotor rehabilitation, showing no difference as to the effect of telerehabilitation compared to other rehabilitative interventions in neurological diseases. Furthermore, within the framework of an EU FP7 project focused on Integrated Home Care, was performed a review on home care in stroke patients, evidencing relevant suggestions to plan telerehabilitation trials, in order to observe the expected effectiveness from a multi-domains point of view in clinical, financial and social perspectives.

A multi-domain Health Technology Assessment approach was set up by the Istituto Superiore di Sanità (ISS), validated and implemented within the EU Project CLEAR. The model, a specialization of EUnet Health Technology Assessment model to telerehabilitation services, was applied to a 960-patients Pilot study in 4 EU Countries to address remote rehabilitation and management of several chronic neurological and motor diseases and was found appropriate for the purpose. The above ISS Health Technology Assessment model proved to have the potential to investigate telerehabilitation services in agreement with the Italian Guidelines on Telemedicine. Highly relevant, it allows exceeding the boundaries and limitations of a specific Hospital-based Health Technology Assessment, thus reaching the more general level of a national-based Health Technology Assessment.

This clinical study with medical device, multicenter, randomized controlled trial with blinded evaluation (single-blind, i.e. the evaluating doctor will be blinded) on cerebral stroke patients, will have the following aims:

Primary objective

• Verify the non-inferiority from the point of view of post-treatment clinical efficacy, in terms of motor, cognitive and language functions, of a "multidomain" telerehabilitation protocol compared to conventional outpatient rehabilitation management in brain stroke patients. The lack of statistically significant differences between the two groups regarding the effects of the treatment for each treated domain will be considered an indication of non-inferiority.

Secondary objectives

* Verify the non-inferiority from the point of view of clinical efficacy 4 weeks after the end of the treatment, in terms of the motor (assessed with Fughl-Meyer assessment), cognitive (Oxford cognitive screen) and language functions (Aachener Aphasia Test), of a "multidomain" telerehabilitation protocol compared to taking charge Conventional outpatient rehabilitation in patients with brain stroke outcomes.
* Compare the effects of a "multidomain" telerehabilitation with a conventional rehabilitation treatment in terms of disability (Barthel Index) and quality of life (Beck Depression Inventory scale, il Short-Form-36 health outcome, la Perceived Disease Impact Scale, la Caregiver Burden Inventory) after post-treatment and 4 weeks after the end of the same.
* Compare a "multidomain" telerehabilitation treatment with a conventional rehabilitation treatment based on an accurate economic analysis in terms of cost-effectiveness, cost-benefit and cost-utility.
* Evaluate the role of "multidomain" telerehabilitation in terms of ease of use, clinical efficacy and cost-effectiveness (Satisfaction Measure Questionnaire, Hospital Readmission Rate, la Service Problem Form e Cost and Time Form) by comparing patients suffering from cerebral stroke results discharged early from the hospital (duration of hospitalization less than 4 weeks) with those discharged after a prolonged hospitalization (duration of hospitalization longer than 4 weeks). In this regard, hospital stay days (stroke units and neurorehabilitation) will be considered.

The inclusion and exclusion criteria are described in the dedicated section, as the description of the outcome measures also.

Once informed consent is obtained for participation in the study, patients will be randomized to conventional rehabilitation therapy or telerehabilitation.

Patients in the telerehabilitation experimental group will undergo 20 sessions (1 hour a day, 5 days a week for 4 consecutive weeks) of "multidomain" telerehabilitation (motor, speech and/or cognitive) with VRRS, K-Wand and Khymu connected to a workstation (Telecockpit):

* VRRS is a medical device to perform cognitive telerehabilitation and home speech therapy in online mode (the therapist connects via a telecockpit with integrated video conference and takes remote control of the device at the patient's home interacting with it in real-time) or offline ( the patient performs the personalized card of exercises, guided by a virtual assistant called "Smart Virtual Assistant" who is able to accompany him interactively in real-time throughout the duration of the rehabilitation treatment session).
* K-Wand is an additional device to VRRS for motor telerehabilitation of the upper limb and trunk. It works with a set of motion sensors through light recognition technology.
* Khymu is a set of sensors added to the VRRS used to carry out motor telerehabilitation activities of the lower limb. The use in combination with the K-Wand is able to allow "full-body" motor telerehabilitation.

Patients will have at their home a special workstation connected to the internet. The same equipment will also be present in the reference structure. As part of the study protocol, only the online telerehabilitation mode will be used, with a direct and bidirectional connection between the two devices, also including an audio and video teleconference. The rehabilitator will be able to remotely control the patient's system: send the exercises necessary for online treatment, check its execution on its own screen, modify them according to clinical needs and monitor the patient's activity thanks to the camera. The patient, in turn, will see on his screen the exercises to be performed, their realization and the results achieved by seeing and listening to the operator who is following him.

For motor treatments, the patient will have to move the end-effector (object or limb) following the trajectory of the corresponding virtual activity displayed on his screen. Cognitive exercises will focus on attentional skills and executive functions.

The rehabilitation of language will be based on exercises of interpretation and production of written and oral words.

With regard to patients assigned to the conventional therapy group, they will undergo 20 sessions (1 hour a day, 5 days a week for 4 consecutive weeks) of "multidomain" rehabilitation (motor, speech and/or cognitive) according to a conventional regime approach outpatient. Currently, it is not possible a priori to precisely define the instruments that will be used during rehabilitation management. These, in fact, will have to be defined on a case-by-case basis on the basis of the physiatric visit and the rehabilitation team's project/intervention program, which is periodically updated to follow the different phases of the patient's clinical evolution. Therefore, the telerehabilitation or conventional treatment methods that will be put in place (the type of therapeutic exercise, the modality of cognitive stimulation and/or taking care of speech therapy) will be determined for each patient on the basis of the needs emerging from the physiatric examination performed at T0, defined according to the Individual Rehabilitation Project and applied according to each Rehabilitation Program (motor, cognitive and/or speech therapy) periodically updated.

Sample size estimation Considering the main outcome measure, the level of functional impairment measured at the FMA, and referring to a Cohen effect-size d of 0.64 calculated on the basis of the data reported on this regard in the literature, telerehabilitation group 53.6 (7.7) and conventional group 49.5 (4.8) [1], given an alpha level of 5%, the two-tailed Mann-Whitney test and a power of 80% (ß), was calculated that a sample size of 82 patients (41 subjects per group) may be sufficient to observe any significant difference between the 2 groups.

Taking into account a possible drop-out rate of about 10%, the sample size was increased by 4 subjects per group, arriving at a final calculation of 90 patients (45 subjects per group) to be enrolled. The calculation was made using the statistical program PASS 14.0.8.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of ischemic brain stroke documented radiologically by brain CT or MRI;
* aphasia documented at the Aachener Aphasia Test (AAT) and/or presence of cognitive deficits documented at the neuropsychological assessment with the Oxford Cognitive Screen (OCS).
* availability of ADSL or higher internet connection at home
* ability of the subject and/or caregiver to understand and use the telerehabilitation system
* signature of informed consent

Exclusion Criteria:

* contemporary participation in other clinical studies;
* cognitive impairment defined as a Montreal Cognitive Assessment (MoCA) score <26;
* bone deformities as a consequence of previous traumatic events in the 4 limbs;
* contractures fixed to the 4 limbs assessed as 4/4 on the modified Ashworth scale (MAS);
* other neurological and orthopaedic diseases interfering with the study.

Particularly vulnerable populations. The following cannot be included in the study:

* patients with judicial interdiction
* patients with supportive administration
* institutionalized patients

Criteria for the ongoing exit from the study

* Relapse of disease during the study period
* Withdrawal of informed consent to participate in the study
* Impossibility to carry out the rehabilitation treatment or the assessments required by the study protocol according to the defined schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Changes at the Fugl-Meyer Assessment score between the time frame | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Fugl-Meyer Assessment allows quantifying the degree of post-stroke disability through the evaluation of the following 5 domains of interest. In the upper and lower limbs: the motor function; sensory function; the range of motion; joint pain. The last domain is balance control. The maximum possible score in the Fugl-Meyer scale is 226, which corresponds to full sensory-motor recovery.
Changes at the Aachener Aphasia Test score between the time frame | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Aachener Aphasia Test for the evaluation of aphasia is composed of 6 sections: spontaneous language, token test, repetition, written language (reading aloud, dictated by composition and dictated by handwriting), denomination (sentences, words, complex words) and oral and written comprehension. All items in the subtests repetition, written language, naming and comprehension are scored on a four-point scale, where 3 represents normal performance and 0 no response, preservation, automatism, or totally unrelated to the target.
Changes at the Oxford Cognitive Screen score between the time frame | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Oxford Cognitive Screen is a short and efficient cognitive screening tool that can be delivered at the bedside in acute stroke. OCS is easy to administer and score and importantly is inclusive for patients with aphasia and neglect. OCS returns a single, not divisible visual snapshot of a patient's cognitive profile, which at a glance demonstrates the specific cognitive domain impairments in Attention, Language, Praxis, Number and Memory.

SECONDARY OUTCOMES:
Barthel Index (BI) | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Barthel Index explores 10 items related to movement, walking, personal hygiene, ability to eat, intestinal and urinary continence.
  The resulting score expresses the degree of assistance that the patient's condition requires in daily activities. The value zero indicates a totally dependent patient, while the value 100, which represents the maximum, indicates a fully autonomous patient.
Beck Depression Inventory scale (BDI-scale) | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  Beck Depression Inventory scale is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The twenty-one questions are about how the subject has been feeling in the last week. Each question has a set of at least four possible responses, ranging in intensity (0 I do not feel sad; 1 I feel sad; 2 I am sad all the time and I can't snap out of it; 3 I am so sad or unhappy that I can't stand it). Higher total scores indicate more severe depressive symptoms.
Short-Form-36 (SF-36) | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  Short Form 36 is a 36-item, patient-reported survey on patient health. The SF-36 is a measure of health status and consists of eight scaled scores (vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role; functioning; social role functioning; mental health) which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Perceived Disease Impact Scale (PDIS) | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The perceived disease impact scale (PDIS) was developed to measure the influence of the illness on various life domains, including well-being, lifestyle, activities, relationships, work, personality, interests and trust in own body.
  It's based on 20 items consisted of a 7-point Likert scale ranging from 'very negatively' (-3) to 'very positively' (+3).
Caregiver Burden Inventory | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Caregiver Burden Inventory comprises 24 closed questions divided into five dimensions: time-dependence, developmental, physical, social and emotional burden. There are five items in each dimension except for physical burden, which has four items dedicated to. Each item is given a score between 0 (not at all descriptive) and 4 (very descriptive), where higher scores indicate greater caregiver burden.
Client Satisfaction Questionnaire | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  The Client Satisfaction Questionnaire is a self-report questionnaire constructed to measure satisfaction with services received by individuals and families. The scales have been broadly adopted, nationally and internationally, by investigators and service program personnel who use the instruments for scientific work, evaluation research, and program planning. Using a logic model, items were drawn from a large pool of items written by Larsen et al. covering nine conceptual domains of client satisfaction: physical surroundings; procedures; support staff; kind or type of service; treatment staff; quality of service; amount, length, or quantity of service; the outcome of service; and general satisfaction. The possible answers are as follow 1=Poor' 2=Fair' 3=Good' 4=Excellent or 1= No' definitely not' 2= No' not really' 3=Yes' generally' 4=Yes' definitely on the base of the questions. The higher the score the greater the satisfaction.
Hospital Readmission Rate | T0 (baseline) - T1 (4 weeks) - T2 (8 weeks)
  A hospital readmission is an episode when a patient who had been discharged from a hospital is admitted again within a specified time (within 8 weeks of discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Universita di Verona
Locations (1):
- Section of Clinical Neurology, Department Neurological, Neuropsychological, Morphological and Movement Sciences, University of Verona, Verona, Italy, Verona, Italy

REFERENCES:
- [Result] Piron L, Turolla A, Agostini M, Zucconi C, Cortese F, Zampolini M, Zannini M, Dam M, Ventura L, Battauz M, Tonin P. Exercises for paretic upper limb after stroke: a combined virtual-reality and telemedicine approach. J Rehabil Med. 2009 Nov;41(12):1016-102. doi: 10.2340/16501977-0459. PMID 19841835